CLINICAL TRIAL: NCT04399902
Title: STudy to ActivelY WARM Trauma Patients (STAY WARM): A Feasibility Pilot Evaluation
Brief Title: Study to Actively Warm Trauma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Luis Teodoro da Luz, Staff Physician, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STAY WARM Trial
Record Dates: First submitted 2020-03-30; First posted 2020-05-22 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Massive Blood Loss; Hypothermia
Keywords: warming blankets; trauma; bleeding
MeSH Terms: conditions — Hypothermia; Wounds and Injuries; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study blanket (Experimental): Two standard warmed hospital blankets will be placed on top of the patient and the study blanket on top of the standard warmed blankets, covering as much of the patient as possible, at the discretion of the care team. At all times, clinicians should ensure that the study blanket does not touch the patient's bare skin.The blanket will remain on the patient through their path of care, and removed from the patient at arrival to the ICU/final phase of care, or if the patient temperature exceeds 38˚C at any point.
  Interventions: Device: Thermal Blanket

INTERVENTIONS:
Device: Thermal Blanket — Ready-Heat 6-Panel Blanket (Military style, manufactured by Techtrade LLC). The 6-panel military-style blanket (86cm x 152 cm, 1.13kg) warms to 40˚C in approximately 15-20 minutes and maintains this temperature for 10 hours.

SUMMARY:
This study evaluates the feasibility of using thermal blankets to actively warm massively bleeding trauma patients at Sunnybrook Health Sciences Centre. It is hypothesized that either full thermal blankets or half thermal blankets will be a feasible intervention to implement for the care of massively bleeding trauma patients.

DETAILED DESCRIPTION:
Hypothermia (core body temperature of <36˚C), is a strong risk factor for mortality and poor outcomes in trauma patients due to its negative hemostatic, cardiovascular, respiratory, and renal effects. Current evidence has reported that massively bleeding hypothermic trauma patients have higher odds of mortality in the first 24 hours of hospital admission, increased length of stay, and increased need for transfusion. Standard hospital blankets are used to passively warm patients through resuscitation and treatment until arrival to the ICU. Interventions such as active heating through thermal blankets should be considered to prevent and treat hypothermia upon arrival of patients than standard warmed hospital blankets to prevent deleterious outcomes in this population.

ELIGIBILITY:
Inclusion Criteria:

* Any trauma patient requiring activation of the massive hemorrhage protocol (life- threatening bleeding situation requiring mobilization of blood bank, laboratory and clinical resources, and anticipated need for at least 4 units of red blood cells immediately and component therapy) during the hours when research staff are available. Normothermic (core body temperature between 36˚C or greater) will also be included, as core body temperature drops once resuscitation is initiated.
* Hypothermic patients (temperature ≤ 35˚C) to whom MHP is NOT activated, when Dr. Luis da Luz/trauma fellow is on call as Trauma Team Leader will also be included.

Exclusion Criteria:

* Patients known to be pregnant
* Patients who die in the trauma bay
* Patients excluded at the discretion of the TTL based on use of the blanket not appearing feasible given the sustained injuries, multiple procedures being conducted in the trauma, or patients who seem to have unsurvivable injuries.
* Patients admitted during study off-hours.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Was the blanket applied to the patient? | Through study completion, an average of 24 hours
  Binary indication of whether or not the blanket is applied to the patient
Were patient temperatures recorded? | Through study completion, an average of 24 hours
  At least 2 temperature recordings (1 in the trauma bay and 1 in the next phase of care - CT scanner suite, angioembolozation suite, emergency department [ED], or operating room), or preferentially, at the final phase of care usually the ICU or ED
Did the blanket remain on the patient? | Through study completion, an average of 24 hours
  Binary indication of whether or not the blanket is kept on the patient in each phase of care until arrival to ICU (1, 2, 3, 4, 5, and 6-hours post initial application of the blanket)

SECONDARY OUTCOMES:
Was the blanket placed directly on the patients skin? | Through study completion, an average of 24 hours
  Number of times blanket is placed directly on the skin
Cold Discomfort Questionnaire | Up to 2 weeks
  Assess cold discomfort of the patient during resuscitation (min value=0 [warm], max value=10 [unbearably cold])
Did the patients temperature exceed 38 degrees Celsius? | Through study completion, an average of 24 hours
  Binary outcome of whether patient temperature exceeded 38 degrees Celsius throughout phases of care
Did the patient experience any redness and/or burns? | Through study completion, an average of 24 hours
  Number of times redness and/or burns are reported by the patient and/or treating clinician

CONTACTS AND LOCATIONS:
Overall Officials: Luis T da Luz, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

REFERENCES:
- [Derived] Strauss R, Kron A, Callum J, Armali C, Modi D, Notario L, D'Empaire PP, Tillmann BW, Pannell D, Tien H, Nathens A, Beckett A, da Luz LT. STudy to ActivelY WARM trauma patients (STAY WARM): a pilot study assessing feasibility of self-warming blankets in patients requiring a massive hemorrhage protocol activation. Eur J Trauma Emerg Surg. 2024 Oct;50(5):2289-2294. doi: 10.1007/s00068-024-02612-w. Epub 2024 Aug 7. PMID 39112757